CLINICAL TRIAL: NCT03477552
Title: Efficacy of AccuVein V400 to Facilitate Peripheral Intravenous Placement in Sickle Cell Disease Adults With Vaso-occlusive Crisis : a Randomized Clinical Trial
Brief Title: Transillumination Device for Peripheral Intravenous Placement in Patients With Sickle Cell Disease (PERFID)
Acronym: PERFID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K160919J; 2017-AO2746-47 (Other Grant/Funding Number: ANSM); PHRIP-16-0139 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2018-02-07; First posted 2018-03-26 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Sickle Cell Crisis
Keywords: Sickle Cell Crisis; intravenous catheter; transillumination
MeSH Terms: conditions — Vaso-Occlusive Crises

STUDY DESIGN:
Intervention Model Description: Adult sickle cell patients who need of a new peripheral intravenous catheter placement (for fluid or porphine therapy) will be randomized between two arms : usual technique or use of the AccuveinV400® device). The randomization list (ratio 1: 1) will be made by the statistician of the study using the SAS software and balanced by random blocks of small size (2, 4, 6) to make it unpredictable. The randomization will be stratified on the center and the number of hospitalizations in the previous year (>3, <3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Accuvein V400 device (Experimental): In the Accuvein group, the nurse uses the Accuvein device to identify the veins before any puncture to infuse the patient and then proceeds as usual, under illumination of the device.
  Interventions: Device: Accuvein V400 device
- Routine procedure (Active Comparator): In the control group, the nurse proceeds as usual to infuse the patient (visual identification in the light of the chamber and palpation)
  Interventions: Other: Routine procedure

INTERVENTIONS:
Device: Accuvein V400 device — Sickle cell patients who need a new vein puncture in order to infuse them will benefit of AccuveinV400 device to illuminate their venous network
  Arms: Accuvein V400 device
Other: Routine procedure — In the control group, the nurse proceeds as usual to infuse the patient (visual identification in the light of the chamber and palpation)
  Arms: Routine procedure

SUMMARY:
The primary goal of this randomized, controlled, open-label study is to determine the efficacy of AccuveinV400 (a transillumination veins device) to facilitate peripheral intravenous (IVP) catheter placement during a vaso-oclusive crisis. The investigators hypothesized that the number of attempts to a successful placement of a peripheral IV, our primary outcome, would be shorter with the assistance of the Accuvein V400. It is also expected that AccuveinV400 will reduce the time of the procedure, the rate of failure, the technique-related pain.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell patients (all genotypes)
* Patients hospitalized for uncomplicated vaso-occlusive crisis (CVO) in Internal/general Medicine department
* Patients requiring the placement or replacement of a peripheral intra-venous catheter in the Department of Internal/general Medicine
* Patients arrived in the internal/general medicine department of the hospital between 9h and 18h and except weekends
* Signed informed consent.
* Affiliated to the French health care insurance.

Exclusion Criteria:

* Signs of shock
* Acute chest Syndrome
* Central venous catheter already present
* Indication to have a central venous catheter from the ourset
* Patient who has already participated to the PERFID study during the current hospitalization
* Refusal of the patient's participation
* Pregnant or lactating woman
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of venipunctures | Time of the infusion procedure
  Number of venipunctures until the peripheral IV placement (with a retrograde blood sample) or before failure (discontinuation after at least 3 attempts by 2 nurses and a maximum of 9 attempts in total).

SECONDARY OUTCOMES:
Time of the procedure | Time of the infusion procedure
  Time from the tourniquet inflation to the insertion of the catheter with a retrograde blood sample was recorded with a chronometer
Procedure failure | Time of the infusion procedure
  Percentage of the procedure failure
The need of a central venous catheter | Time of the infusion procedure
  Percentage of use of a central venous catheter due to failure of peripheral perfusion.
Patient bone pain before and after the procedure | Before and within 1 hour after a successful peripheral IV placement
  Patient bone pain will be evaluated by Visual Analogue Scale (between 0=no pain to10=intolerable pain) before and after the infusion procedure
Anxiety before and after the procedure | Just before and within 1 hour after a successful peripheral IV placement
  Patient and nurse anxiety will be evaluated by a visual 5 points-Likert scale (between 1=not at all anxiety to 5=extremely anxious) of anxiety before and after the procedure
Patient satisfaction (pain) | Within 1 hour after a successful peripheral IV placement
  Patient pain related to the procedure will be evaluated by Visual Analogue Scale (between 0=no pain to10=intolerable pain)
Patient satisfaction (procedure) | Within 1 hour after a successful peripheral IV placement
  Patient satisfaction of the procedure will be evaluated by a visual 5-points Likert scale (between 1=not at all anxiety to 5=extremely anxious) of satisfaction of the procedure
Nurse satisfaction (procedure) | Within 1 hour after a successful peripheral IV placement
  Nurse global satisfaction of the procedure will be evaluated by Likert scale (between 1=not at all anxiety to 5=extremely anxious)
Nurse satisfaction (quality of placement) | Within 1 hour after a successful peripheral IV placement
  Nurse satisfaction of the quality of the peripheral intravenous placement will be evaluated by Likert scale (between 1=not at all anxiety to 5=extremely anxious)
Qualitative interview of the Accuvein use | An average of one week after the procedure
  Verbatim of a semi-structured interview by a psychologist of 10 to 15 patients (and their nurse) often hospitalized, in the Accuvein Arm
Side effects of the procedure | Time of the infusion procedure
  Complication rate of the peripheral venous catheter procedure (hematoma, bleeding, malaise).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Benoit Arlet, MD,PhD, Principal Investigator — Medicine interne department, Europeen Georges Pompidou Hopital, Paris, France; Eric Fischer, Principal Investigator — Medicine interne department, Europeen Georges Pompidou Hospital, Paris, France; François Lionnet, MD, Principal Investigator — Medicine interne department, Tenon Hospital, Paris, France
Locations (2):
- France (2):
  - CHU H. Mondor, Créteil
  - AP-HP - Hopital Europeen Georges-Pompidou Paris, France, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corbasson A, Fischer E, Vilfaillot A, Da Costa AB, Charmettan M, Ferreira M, Barthelemy C, Namaoui W, Khimoud D, Beaudoin A, Berkani L, Guillaud C, Khellaf M, Flamarion E, Michon A, Lafont E, Cheminet G, Chatellier G, Pouchot J, Ranque B, Arlet JB. Efficacy of a vein visualisation device for facilitating peripheral venous line placement in adult patients with sickle cell disease: A randomised clinical trial. Int J Nurs Stud. 2025 Mar;163:104988. doi: 10.1016/j.ijnurstu.2024.104988. Epub 2024 Dec 19. PMID 39787687